CLINICAL TRIAL: NCT05787769
Title: A Randomized Trial to Evaluate Efficacy and Safety of Intracavernosal Injection of Platelet-Rich Plasma Versus Phosphodiesterase Type-5 Inhibitors for Treatment of Erectile Dysfunction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP-ED
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Erectile Dysfunction Following Radiation Therapy; Phosphodiesterase Inhibitor Adverse Reaction; Platelet- Rich Plasma (PRP)
Keywords: Erectile Dysfunction , Phosphodiesterase Inhibitor Adverse Reaction, platelet- rich plasma
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P shot arm (Active Comparator): Drug: Autologous Platelet Rich Plasma + placebo tab Each injection session will consist of a total of 10 mL PRP infused slowly over a 2-minute period; 5 mL each injected to the right and left corpus cavernosum.
  Interventions: Drug: P shot arm ( Autologous Platelet Rich Plasma)
- PDE5i arm (Active Comparator): Drug: Tadalafil + placebo injection Patients will be treated by tadalafil 5 mg tablet daily in addition to four Tadalafil 5 mg tablet 3 hours before intercourse on demand in addition to placebo injection. Each injection session will consist of a total of 10 mL saline solution infused slowly over a 2-minute period; 5 mL each injected to the right and left corpus cavernosum.
  Interventions: Drug: PDE5i arm

INTERVENTIONS:
Drug: P shot arm ( Autologous Platelet Rich Plasma) — Autologous Platelet Rich Plasma + placebo tab Each injection session will consist of a total of 10 mL PRP infused slowly over a 2-minute period; 5 mL each injected to the right and left corpus cavernosum
  Other Names: Autologous Platelet Rich Plasma
  Arms: P shot arm
Drug: PDE5i arm — Patients will be treated by tadalafil 5 mg tablet daily in addition to four Tadalafil 5 mg tablet 3 hours before intercourse on demand in addition to placebo injection. Each injection session will consist of a total of 10 mL saline solution infused slowly over a 2-minute period; 5 mL each injected to the right and left corpus cavernosum.
  Arms: PDE5i arm

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of intracavernosal injection of PRP in patients with moderate to severe ED.

ELIGIBILITY:
Inclusion Criteria:

* 1) Signed an ethics committee-reviewed and approved informed consent form. 2) Subjects must meet all inclusion criteria to be eligible for study enrollment.

  3) Men between 30 and 75 years old, 4) Sexually active in a stable, heterosexual relationship of at least six months duration.

  5) ED for at least 6 months with an IIEF-EF between 5 and 16 points, inclusive. 6) ED of vascular origin. 7) Subjects agree to attempt vaginal intercourse at least 4 times every month after the end of the treatment and agree to document the outcome using the Sexual Encounter Profile (SEP) and the Erection Hardness Score (EHS).

  8) Commitment not to use other treatment for ED during the study (herbal, topical, intraurethral, intracavernosal, etc.).

  9) Willingness and ability to comply with study procedures, other measurements instruments and visit schedules and able to follow oral and written instructions.

Exclusion Criteria:

* 1) Refuse to complete study requirements. 2) Psychogenic ED as determined by study investigator. 3) ED of neurogenic origin (radical cystectomy, radical prostatectomy, pelvic surgery, spinal cord injury, multiple sclerosis, DM is not included unless documented diabetic neuropathy).

  4) Previous penile surgery of any kind (except circumcision, frenuloplasty and condyloma removal), such as penile prosthesis, penile lengthening, penile cancer surgery, penile plication, grafting.

  5) Previous history of penile fracture, Peyronie's disease or priapism. 6) Previous radiation to pelvis. 7) History of symptomatic hypogonadism (testosterone level <346ng/dl) not treated.

  8) Major hematologic, renal, or hepatic abnormalities. 9) Severe decompensated cardiac, CNS or vascular insufficiency. 10) Poorly controlled hypertension or DM (HbA1c >12%). 11) Neoplasm of any origin in active treatment or active progression or recovering from cancer within 12 months prior to enrollment.

  12) History of alcohol abuse or drug. 13) Treatment with oral anticoagulants, antiandrogens or nitrates. 14) Thrombopenia less than 100 x 103 / L. 15) Hemoglobin <10g/dl. 16) Poor venous access or any other circumstance that preclude an apheresis procedure.

  17) Sexually inactive in recent months. 18) participation in another study that may interfere with the results or conclusions of this study.

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-25 (Estimated); Study Completion 2025-01-25 (Estimated)

PRIMARY OUTCOMES:
efficacy of intracavernosal injections of platelet-rich plasma (PRP) in patients Erectile Dysfunction. | 6 months
  assessed by the proportion of patients attaining minimal clinically important difference in the international index of erectile function - erection dpmain.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-assmy, Study Director — Mansoura University
Locations (1):
- Mansoura urology and nephrology center, Al Mansurah, Outside U.S./Canada, Egypt